CLINICAL TRIAL: NCT02747277
Title: Analysis of B Cells From Autoimmune Individuals
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-0541; UL1TR001082 (NIH)
Record Dates: First submitted 2016-04-14; First posted 2016-04-21 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Lupus Erythematosus; Rheumatoid Arthritis; Type 1 Diabetes
MeSH Terms: conditions — Arthritis, Rheumatoid; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, umbilical cord blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study aims at finding out if individual with autoimmunity exhibit increased numbers of B cells that express two types (instead of one type) of antibodies, and if B cells of individuals genetically susceptible to autoimmunity display defects in the biological process of tolerance, which removes B cells that participate in autoimmunity.

DETAILED DESCRIPTION:
Peripheral blood B cells of SLE patients are analyzed by flow cytometry to determine the frequency of B cells co-expressing immunoglobulin kappa an lambda light chains. This frequency is correlated to the disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult Males and Females diagnosed with Lupus;
* Adult Females who are pregnant and diagnosed with:

  * lupus erythematosus
  * rheumatoid arthritis, or
  * type 1 diabetes.

Exclusion Criteria:

* Adult males or adult females treated with B-cell depletion therapies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females with a diagnoses of lupus erythematosus, rheumatoid arthritis, or type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-05; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Frequency of kappa to lambda ratios of B cells in blood of autoimmune adults | 1 day
  For peripheral adult blood, the main outcome measure is the frequency of κ/λ (kappa to lambda ratios) dual immunoglobulin B cells within the overall B (CD19+ or CD20+) cell population. The collected data will be aggregated as the average frequency of κ/λ B cells in subjects with autoimmunity relative to healthy controls.
Frequency of CD19 and IgM low B cells in cord blood of babies born from autoimmune mothers | 1 day
  For cord blood samples, the main outcome measurement is the frequency of B cells that express both low levels of CD19 and IgM within the total (CD19+ or CD20+) B cell population. The collected data will be aggregated as the average frequency of CD19low/IgMlow B cells in subjects that were born from autoimmune mothers relative to those born from healthy mothers. Moreover, data will also be stratified in respect to the presence or absence of the PTPN22-R620W allele, which is a risk allele for autoimmunity.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Pelanda, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data will be presented at conferences and eventually published in peer-reviewed publication.

REFERENCES:
- [Result] Peterson JN, Boackle SA, Taitano SH, Sang A, Lang J, Kelly M, Rahkola JT, Miranda AM, Sheridan RM, Thurman JM, Rao VK, Torres RM, Pelanda R. Elevated Detection of Dual Antibody B Cells Identifies Lupus Patients With B Cell-Reactive VH4-34 Autoantibodies. Front Immunol. 2022 Feb 4;13:795209. doi: 10.3389/fimmu.2022.795209. eCollection 2022. PMID 35185888
- [Result] Alves da Costa T, Peterson JN, Lang J, Shulman J, Liang X, Freed BM, Boackle SA, Lauzurica P, Torres RM, Pelanda R. Central human B cell tolerance manifests with a distinctive cell phenotype and is enforced via CXCR4 signaling in hu-mice. Proc Natl Acad Sci U S A. 2021 Apr 20;118(16):e2021570118. doi: 10.1073/pnas.2021570118. PMID 33850015